CLINICAL TRIAL: NCT03533881
Title: Evaluation of Metabolic Effects and in Modulation of Food Behaviour of Arom Digest Slim Product in Association With Minimal Nutritional Changes in Overweight Patients
Brief Title: Effects of Arom Digest Slim on Metabolic Profile and Food Behaviour in Overweight Persons
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SC Aromaarmony SRL (Industry)
Responsible Party: Principal Investigator, Monica Goia-Socol, Assist. Prof. Dr. Monica Goia-Socol, MD, PhD, SC Aromaarmony SRL
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Arom Digest Slim
Record Dates: First submitted 2018-04-25; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Metabolic Syndrome
Keywords: collagen; volatile oils; metabolic syndrome; insulin resistance
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Group 1: following minimal nutritional changes Group 2: following minimal nutritional changes and taking Arom Digest Slim
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arom Digest Slim and nutritional changes (Active Comparator): Subjects take collagen and follow minimal nutritional changes.
  Interventions: Dietary Supplement: Arom Digest Slim; Behavioral: Nutritional changes
- Nutritional changes (Active Comparator): Subjects only follow minimal nutritional changes
  Interventions: Behavioral: Nutritional changes

INTERVENTIONS:
Dietary Supplement: Arom Digest Slim — Arom Digest Slim is a dietary supplement approved in Romania by SNPMAPS, with notification number AA 10802/2017.
  It contains: hydrolyzed fish collagen (94,8 %) and volatile oils (5,2 %): Citrus paradisi (2,40 %), Citrus aurantifolia (1,24 %), Menta avensis (0,92 %), Cinamomum zeylanicum (0,56%) Patients take 4 grams of supplement per day; the supplement is dissolved in 750 ml water and drunk throughout the day
  Arms: Arom Digest Slim and nutritional changes
Behavioral: Nutritional changes — Education to increase the fruits and vegetables, decrease refined carbohydrates, decrease high fat animal products, regulation of meal programme, increase water intake to at least 1,5 liters per day

SUMMARY:
The present study aims to evaluate the efficacy of Arom Digest Slim in facilitating weight reduction along with a series of minimal nutritional interventions.

DETAILED DESCRIPTION:
Arom Digest Slim is a blend of fish collagen and essential oils. It will be administered in a group of overweight females wich also undertake minimal nutritional changes. The group will be compared with a group following only minimal nutritional changes.

ELIGIBILITY:
Inclusion Criteria:

* females 18 to 60 years old

Exclusion Criteria:

* cardiovascular, psychiatric and neurologic chronic conditions and medication
* acute conditions
* patients with hypersensitivity to any components of the product

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-02-15 (Estimated); Study Completion 2019-04-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Insulin Resistance index (HOMA) at 60 days (Biochemical assessment) | baseline and 60 days
  calculated from serum level of glucose and insulin: HOMA-IR = (insulin (µU/mL) x glycemia (mg/dL))/405
Change from Baseline Lipids at 60 days (Biochemical assessment) | baseline and 60 days
  total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides - serum level (mg/dl)
Change from Baseline Food behavior at 60 days (Three Factor Eating Questionnaire 18 (TEFQ 18)) | baseline and 60 days
  Food behavior questionnaire: Three Factor Eating Questionnaire 18 (TEFQ 18)
  Assessed parameters:
  Uncontrolled eating - minimal possible value 9, maximal possible value 54 points Cognitive restriction - minimal possible value 3, maximal possible value 12 points Emotional eating - minimal possible value 5, maximal possible value 24 points Higher values represent a worse outcome. Subscales are summed to compute a total score.
Change from Baseline Bioimpedance parameters at 60 days (measured using InBody720 equipment) | baseline and 60 days
  Bioimpedance using InBody720 equipment (Biospace Co., Ltd.)
  Assessed parameters:
  A. Body Composition Analysis (9 items): Intracellular Water, Extracellular Water, Protein Mass (kg), Mineral Mass (kg), Body Fat Mass (kg), Total Body Water, Soft Lean Mass (kg), Fat Free Mass (kg), Weight (kg) B. Muscle-Fat Analysis(3 items): Weight (kg), Skeletal Muscle Mass (kg), Body Fat Mass (kg) C. Obesity Diagnosis: Body Mass Index(BMI, kg/m2), Percent Body Fat (%), Waist-Hip Ratio D. Lean Balance (5 items): Right Arm (kg), Left Arm (kg), Trunk (kg), Right Leg (kg), Left Leg (kg) E. Visceral Fat Area: Norma l<100cm2 Over : 100~150cm2 Extremely over : >150cm2 F. Weight Control(4 items): Target Weight (kg), Weight Control(kg), Fat Control(kg), Muscle Control(kg) F. Fitness Score: The Fitness Score is an arbitrary score based on the measured muscle and fat mass for the motivation of the subjects. Under 70 : Weak Type 70~90 : NormalType Over 90 : Athletic Type

CONTACTS AND LOCATIONS:
Overall Officials: Monica Goia-Socol, MD, PhD, Principal Investigator — Endocrinology Department, University of Medicine and Pharmacy Cluj-Napoca, Romania
Locations (1):
- Endocrinology Department, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee EJ, Hur J, Ham SA, Jo Y, Lee S, Choi MJ, Seo HG. Fish collagen peptide inhibits the adipogenic differentiation of preadipocytes and ameliorates obesity in high fat diet-fed mice. Int J Biol Macromol. 2017 Nov;104(Pt A):281-286. doi: 10.1016/j.ijbiomac.2017.05.151. Epub 2017 Jun 9. PMID 28602994
- [Background] Subhan F, Kang HY, Lim Y, Ikram M, Baek SY, Jin S, Jeong YH, Kwak JY, Yoon S. Fish Scale Collagen Peptides Protect against CoCl2/TNF-alpha-Induced Cytotoxicity and Inflammation via Inhibition of ROS, MAPK, and NF-kappaB Pathways in HaCaT Cells. Oxid Med Cell Longev. 2017;2017:9703609. doi: 10.1155/2017/9703609. Epub 2017 Jun 22. PMID 28717410
- [Background] Lone J, Yun JW. Monoterpene limonene induces brown fat-like phenotype in 3T3-L1 white adipocytes. Life Sci. 2016 May 15;153:198-206. doi: 10.1016/j.lfs.2016.04.010. Epub 2016 Apr 9. PMID 27071835
- [Background] Medagama AB. The glycaemic outcomes of Cinnamon, a review of the experimental evidence and clinical trials. Nutr J. 2015 Oct 16;14:108. doi: 10.1186/s12937-015-0098-9. PMID 26475130
- [Background] Maenner K, Vahjen W, Simon O. Studies on the effects of essential-oil-based feed additives on performance, ileal nutrient digestibility, and selected bacterial groups in the gastrointestinal tract of piglets. J Anim Sci. 2011 Jul;89(7):2106-12. doi: 10.2527/jas.2010-2950. Epub 2011 Feb 25. PMID 21357448
- [Background] Boschi V, Iorio D, Margiotta N, D'Orsi P, Falconi C. The three-factor eating questionnaire in the evaluation of eating behaviour in subjects seeking participation in a dietotherapy programme. Ann Nutr Metab. 2001;45(2):72-7. doi: 10.1159/000046709. PMID 11359032